CLINICAL TRIAL: NCT06863896
Title: Laparoscopic Hartmann's Reversal Procedure ( LHarSal Study)
Brief Title: Laparoscopic Hartmann's Reversal Procedure: In the Absence of Standardized Guidelines, we Started a Database of Patient Submitted Reversal Hartman With Standard Technique and Laparoscopic Technique, Prospectively for One Year and a Follow-up Period of 6 Months
Acronym: LHarSAL
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda USL Toscana Centro (Other)
Responsible Party: Principal Investigator, Carla Vaccaro, Principal Investigator Carla Vaccaro, Azienda USL Toscana Centro
Other Study IDs: v 1.0 del 01/01/2025
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Colostomy - Stoma
Keywords: colostomy; hartmann

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing Reversal Hartmann's procedure with open or laparoscopic technique: The study population includes all consecutive adult patients (≥18 years of age) underwent Hartmann's reversal procedure (open or laparoscopic procedure) in the participating centers
  Interventions: Procedure: Hartmann's reversal

INTERVENTIONS:
Procedure: Hartmann's reversal — Colostomy reversal with laparoscopic technique after Hartmann's procedure ( procto-sigmoidectomy with end colostomy)

SUMMARY:
Several studies have shown laparoscopic technique's advantages, including more rapid post-operative recovery, less post-operative pain, earlier restoration of bowel function, more rapid return to normal diet, and reduced morbidity but it could still remain a complicated operation due to adhesions and difficulty in identifying the rectal stump. Nevertheless, nowadays laparoscopic technique has largely become part of clinical practice even for younger surgeons. Assumed this, and in the lack of prospective studies, we aimed to confirm the advantages of laparoscopic Hartmann reversal (LHR) by confirming the difference in peri-operative outcomes and postoperative complications.

In clinical practice, the first question to be asked is whether there is a right timing for a patient to undergo Hartmann's reversal procedure and whether timing influences the incidence of complications (short-terms and long-terms outcomes). Another aim of the study is to investigate if the length of rectal stump influences the outcome of Hartmann's reversal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, ≥ 18 years old.
2. Patients who underwent Hartmann procedure for diverticulitis, intestinal ischemia or trauma
3. Patients who may face a one-year follow-up.
4. Patients fit for surgery.

Exclusion Criteria:

1. age < 18.
2. patients that have undergone Hartmann's procedure for cancer and also post-Hartmann adjuvant radiotherapy or residual neoplastic disease.
3. immunodepression condition (patients undergoing chemo-radiotherapy and/or immunotherapy, patients undergoing immunosuppressive therapy for autoimmune diseases or transplants, cirrhotic class C and D patients, patients with chronic renal failure undergoing dialysis treatment.)
4. patients with missing data
5. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes all consecutive adult patients (≥18 years of age) underwent Hartmann's reversal procedure (open or laparoscopic procedure) in the participating centers. The decision to perform HR is based on the patients' preference and the attending surgeons' opinion and experience, after evaluating their clinical condition.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
average post-operative hospital stay | from the day of surgery to the the day of discharge from the hospital ( up to 10 days)

IPD SHARING:
Plan to Share IPD: Yes
Primary outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code